CLINICAL TRIAL: NCT02214238
Title: Evaluation of Treatment Efficacy and Comfort of a Modified Positive Airway Pressure Device to Treat Obstructive Sleep Apnea, in Comparison to a Market Released Device.
Brief Title: Evaluation of Treatment Efficacy and Comfort of a Modified Positive Airway Pressure Device to Treat Obstructive Sleep Apnea.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CIA-116
Record Dates: First submitted 2014-08-10; First posted 2014-08-12 (Estimated); Results first posted 2017-04-24 (Actual); Last update posted 2017-04-24 (Actual); Status verified 2017-03

CONDITIONS: Obstructive Sleep Apnea (OSA)
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Market released PAP device (Active Comparator): Use of a market released PAP device
  Interventions: Device: PAP device
- Modified PAP device (Experimental): Us of the modified PAP device
  Interventions: Device: PAP device

INTERVENTIONS:
Device: PAP device

SUMMARY:
This study will test the hypothesis that the modified positive airway pressure (PAP) device for OSA will be no worse than a market released product in terms of its treatment efficacy, comfort and patient compliance. Patients will have their treatment pressure titrated using polysomnography (PSG) in the sleep laboratory, and then in a random order will spend additional time undergoing PSG using both devices, and using both devices at home for 3 weeks. Data will be collected from the PSG studies, device downloads, independent pressure-flow loggers, and custom questionnaires.

DETAILED DESCRIPTION:
The study will be held in two parts. The main portion of the study which compares the modified PAP device and the market released product including the laboratory testing and home testing of the devices will be called 'Part A'. Additional nights using the PAP device with PSG monitoring will be used to gather additional observational flow data to allow distortion testing and investigation of the FPH (Fisher & Paykel Healthcare) SensAwake (an unique feature which automatically lowers the pressure when a patient wakes up) algorithm while using PAP, this is part B.

Part A After the patient has undergone informed consent, their demographic and clinical variables will be collected and entered into a case report form (CRF) before any setup procedure is started. The patient will be asked to complete questionnaires regarding their normal therapy (ESS (Epworth Sleepiness Score), FOSQ (Functional Outcomes of Sleep Questionnaire), custom therapy comfort questionnaire), and then will be set up for a standard PSG. The patient will use their prescribed mask and a clean water chamber and breathing tube which will be connected to the modified PAP device. The patients will sleep on the device throughout the night while having their PAP titrated by a qualified sleep technician. Pressure titration is necessary for two reasons: firstly, it may have been a period of time since the participants last titration, and secondly this version of PAP involves the use of different levels of pressure. Pressures will be titrated according to the AASM (American Academy of Sleep Medicine) Clinical Guidelines for the Manual Titration of Positive Airway Pressure in Patients with OSA.

The participant will be randomized to either the modified PAP or market released device group. They will be issued with a PAP device and a pressure-flow logger to be used at home in the usual manner of their PAP therapy for 3 weeks (+/- 4 days), after which participants will return to the FPH sleep laboratory to participate in a overnight PSG study using their first device. At this visit the participant will also swap to the second PAP device; and the above home use repeated on device 2.

Part B After informed consent form the patient will be set up for a standard PSG, and sleep overnight using the modified PAP device, their prescribed mask, and a clean water chamber and breathing tube. This testing will be performed to provide additional flow data to the development engineers. This includes, but is not limited to, distortion testing and adjustment of device parameters during the sleep study. Distortion testing analyses the impact of the PAP pressure changes on the participants breathing or airflow.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18+
* Diagnosed with OSA by a practicing sleep physician

Exclusion Criteria:

* Patients with a known history of Cerebrospinal fluid leak, abnormalities of the cribriform plate, head trauma and/or pneumocephalus
* Patients with pathologically low blood pressure, pneumothorax, a previous history of pneumothorax, or dehydration.
* Patient with bypassed upper airway
* Other significant sleep disorder(s) (e.g. periodic leg movements, insomnia, central sleep apnea)
* Previous use of a bi-level device with-in the last 2 years (from enrolment date).
* Patients with respiratory failure, bullous lung disease or COPD (Chronic Obstructive Pulmonary Disease).
* Patients with obesity hypoventilation syndrome or congestive heart failure
* Patients that require supplemental oxygen with their CPAP (Continuous Positive Airway Pressure) device
* Patients with implanted or life-supporting electronic medical devices (e.g. cardiac pacemakers)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2014-08; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hanie Yee, Study Director — Fisher & Paykel Healthcare
Locations (1):
- Fisher & Paykel Healthcare, Auckland, New Zealand

RESULTS

PARTICIPANT FLOW:
Groups:
- Market Released PAP Device First, Then Modified PAP Device: Use of a market released PAP device first for 3 week (with a 4 day window) followed by an in lab sleep study. Patient then crossed over to use the modified PAP device for 3 weeks (with a 4 day window) followed by another in lab sleep study.
- Modified PAP Device First, Then Market Released PAP Device: Use of the modified PAP device first for 3 week (with a 4 day window) followed by an in lab sleep study. Patient then crossed over to use the market released PAP device for 3 weeks (with a 4 day window) followed by another in lab sleep study.
Period: Overall Study
Arm/Group | Market Released PAP Device First, Then Modified PAP Device | Modified PAP Device First, Then Market Released PAP Device
Started | 26 | 23
Completed | 20 | 17
Not Completed | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Modified PAP Device First, Then Market Released PAP Device: Us of the modified PAP device first for 3 week (with a 4 day window) followed by an in lab sleep study. Patient then crossed over to use the market released PAP device for 3 weeks (with a 4 day window) followed by another in lab sleep study.
- Total: Total of all reporting groups
Arm/Group | Market Released PAP Device First, Then Modified PAP Device | Modified PAP Device First, Then Market Released PAP Device | Total
Number analyzed (Participants) | 26 | 23 | 49
Age, Continuous [Mean (Full Range); unit: years] | 63.2 [48 to 81] | 58.7 [32 to 81] | 60.9 [32 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 24 | 22 | 46
Region of Enrollment [Number; unit: participants]
  New Zealand | 26 | 23 | 49

OUTCOME MEASURES:

1. Primary Outcome: PAP Treatment Efficacy
Description: The participants apnea hypopnea index (AHI) will be assessed using the PSG data, device download data and the independent pressure-flow logger. The apnea-hypopnea index is the total number of sleep disordered breathing events divided by total sleep time.
Time Frame: After 1 night in the sleep lab and 3 weeks use of the device in the home.
Population: The overall number of participants analyzed is represented independent to which arm the participant started. Out of 49 total patients at baseline, 37 had usable data for analysis after using each device. AHI was compared between devices independent of which order the participants used each device.
Measure: Mean (Standard Deviation); unit: Events per hour
Groups:
- Market Released PAP Device: Use of a market released PAP device
  PAP device
- Modified PAP Device: Use of the modified PAP device
  PAP device
Arm/Group | Market Released PAP Device | Modified PAP Device
Number analyzed (Participants) | 37 | 37
Events per hour | 4.2 (1.0) | 4.0 (1.0)

2. Secondary Outcome: PAP Treatment Comfort
Description: Participants will be administered comfort questionnaires regarding the comfort of all devices. The range of responses is 1 to 5 with 1 being very uncomfortable to 5 being very comfortable.
Time Frame: After 1 night in the sleep lab and 3 weeks use of the device in the home.
Population: The overall number of participants analyzed is represented independent to which arm the participant started. Out of 49 total patients at baseline, 35 had usable data for analysis after using each device. PAP treatment comfort was compared between devices independent of which order the participants used each device.
Measure: Median (Full Range); unit: Units on a Scale
Arm/Group | Market Released PAP Device | Modified PAP Device
Number analyzed (Participants) | 35 | 35
Units on a Scale | 5 [1 to 5] | 5 [1 to 5]

3. Secondary Outcome: PAP Compliance
Description: Participants therapy utilisation will be compared between the two devices using the device data download, and the independent pressure-flow logger.
Time Frame: After 1 night in the sleep lab and 3 weeks use of the device in the home.
Population: The overall number of participants analyzed is represented independent to which arm the participant started. Out of 49 total patients at baseline, 31 had usable data for analysis after using both devices. Compliance was compared between devices independent of which order the participants used each device.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Market Released PAP Device | Modified PAP Device
Number analyzed (Participants) | 31 | 31
Minutes | 438 (13) | 430 (12)

ADVERSE EVENTS:
Time Frame: 6 Weeks
Groups:
- Modified PAP Device: Use of a modified PAP device for 3 more weeks.
- Market Released PAP Device: Use of a market released PAP device for 3 more weeks.
Arm/Group | Modified PAP Device | Market Released PAP Device
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/43
Other Adverse Events (participants affected / at risk) | 5/49 | 3/43
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Modified PAP Device (N=49) | Market Released PAP Device (N=43)
Snoring and somnolence (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nose bleed (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Angioedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Determined by hospital physicians to be related to patients Blood Pressure medications
High AHI on PSG (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Shoulder Operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Ectopic Beats (Cardiac disorders) | 1 (1) | 0 (0) — Observed during PSG
Cricopharyngeal Spasm (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Sensation of lump in the throat

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes